CLINICAL TRIAL: NCT02843100
Title: Modified Exclusive Enteral Nutrition With the Crohn's Disease Exclusion Diet for Induction and Maintenance of Remission and Re-biosis
Brief Title: Diet for Induction and Maintenance of Remission and Re-biosis in Crohn's Disease
Acronym: DIETOMICS-CD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prof. Arie Levine (Other Government)
Responsible Party: Sponsor-Investigator, Prof. Arie Levine, Director, Pediatric Gastroenterology and Nutrition unit, Wolfson Medical Center
Organization: Wolfson Medical Center (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0075-16 WOMC
Record Dates: First submitted 2016-06-22; First posted 2016-07-25 (Estimated); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Crohn's Disease
Keywords: Crohn's Disease; Pediatric; Exclusive Enteral Nutrition; Diet; Microbiome
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Modified Exclusive Enteral Nutrition including two weeks of Exclusive Enteral Nutrition (EEN) using Modulen followed by Partial Enteral Nutrition (PEN) along with the Crohn's Disease Exclusion Diet (CDED) phases 2 & 3 for 24 weeks
  Interventions: Other: Modified Exclusive Enteral Nutrition; Other: Crohn's Disease Exclusion Diet; Other: Partial Enteral Nutrition
- Group 2 (Active Comparator): Standard Exclusive Enteral Nutrition for 8 weeks using Modulen, followed by free diet with gradual reduction of Modulen to 25% of energy needs by week 24.
  Interventions: Other: Partial Enteral Nutrition; Other: Standard Exclusive Enteral Nutrition

INTERVENTIONS:
Other: Modified Exclusive Enteral Nutrition — Two weeks of Exclusive Enteral Nutrition with Modulen
  Other Names: Modulen, Nestle
  Arms: Group 1
Other: Crohn's Disease Exclusion Diet — a limited whole food diet
  Other Names: CDED
  Arms: Group 1
Other: Partial Enteral Nutrition — 25-50% of Energy from formula
  Other Names: Modulen, Nestle
Other: Standard Exclusive Enteral Nutrition — 8 weeks of Exclusive Enteral Nutrition
  Other Names: Modulen, Nestle
  Arms: Group 2

SUMMARY:
The modified-Exclusive Enteral Nutrition (mEEN) is an open label randomized controlled trial in mild to severe Crohn's Disease patients. The purpose of this study is to determine whether induction of remission and maintenance of remission can be achieved with a new dietary strategy that involves only 2 weeks of Exclusive Enteral Nutrition (EEN) with Modulen and 12 weeks of an exclusion diet involving selected table foods. This novel approach will be compared to the gold standard dietary regime involving 8 weeks of EEN.

DETAILED DESCRIPTION:
Rational: Exclusive enteral nutrition (EEN) is an established but difficult to perform method for induction of remission and cannot be used for maintenance of remission. It entails drinking only liquid formula for 8 weeks. Refusal to use or to adhere to this therapy is not uncommon and leads to use of other non- dietary strategies in children including steroids and immunosuppression. The Crohn's Disease Exclusion Diet (CDED) with partial enteral nutrition has been shown to be effective for children with mild to moderate disease. The investigators have developed a maintenance strategy using the CDED.

Objectives: To prove that induction of remission and maintenance of remission can be achieved with a new dietary strategy that involves only 2 weeks of EEN with Modulen and 12 weeks of an exclusion diet involving selected table foods.

Methods: Open label randomized controlled pilot trial comparing two weeks of EEN followed by the CDED and Partial Enteral Nutrition (PEN), to 8 weeks of EEN followed by PEN with free diet. The study will include a control group of healthy children for microbiome studies.

Population: Age 8-18 years with mild to severe active Crohn's disease defined as 15≤Pediatric Crohn's Disease Activity Index (PCDAI)<47.5.

Time frame: The induction of remission phase will last 8 weeks followed by maintenance phase for a period of 24 weeks.

Expected outcomes and significance: If this method proves to be equivalent to EEN, the duration of use of EEN will be only two weeks, allowing more patients access to dietary therapy. More importantly, this study will also evaluate two maintenance strategies and will be the first to evaluate re-biosis.

ELIGIBILITY:
Inclusion criteria:

1. Established diagnosis of Crohn's disease.
2. Patients with mild to severe active Crohn's disease (15≤PCDAI≤47.5)
3. Ages 8-18
4. Duration of disease ≤ 36 months
5. Active inflammation (CRP≥>0.6 mg /dL or ESR≥>20 or Calprotectin≥>200 mcg/gr within the past 3 weeks) during screening
6. Patients with B1, P0 uncomplicated disease at enrollment
7. Patients with disease defined as L1, L4, L3 or L2 limited to cecum, ascending or transverse colon or L2 with left sided disease with terminal ileum or small bowel involvement in the past by the Paris classification (patients with macroscopic disease)
8. Signed informed consent

Exclusion Criteria:

1. Patients with very mild disease (PCDAI 12.5 -15) or very severe disease (PCDAI >47.5)
2. Pregnancy
3. Patients who have disease confined to the colon involving the descending colon, rectum or sigmoid colon and no prior history of small bowel involvement
4. Patients who have active extra intestinal disease (such as Arthritis, Uveitis, Pyoderma Gangrenosum, Erythema Nodosum etc.)
5. Patients with complicated disease (B2, B3)
6. Patients who recently onset use of an immunomodulator <8 weeks, or dose change in past 8 weeks.
7. Patients with current use of biologics, or use in last 8 weeks or current use of systemic steroids
8. Patients who have active perianal disease ( active fistula or abscess)
9. Patients who have positive stool cultures with relevant pathogens,, or positive tests for parasites or C. difficile. Stool tests are mandatory only if diarrhea is present.
10. Patients with fever > 38.3
11. Documented milk protein allergy

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 63 (Actual)
Dates: Start 2018-04-10 (Actual); Primary Completion 2022-05-29 (Actual); Study Completion 2022-05-29 (Actual)

PRIMARY OUTCOMES:
ITT, steroid free Clinical remission (defined as Pediatric Crohn's Disease Activity Index (PCDAI)<10) at week 14 | week 14
  Sustained remission with EEN Vs CDED+PEN

SECONDARY OUTCOMES:
ITT steroid free remission at week 8 | week 8
  Induction of remission
Microbiome composition difference between groups at week 14 | week 14
  Assessment of microbiome composition and metabolomics
3. Reduction of at least 50% from baseline in fecal calprotectin at week 24 for patients on original treatment | week 24
  Mucosal healing assessment
Steroid and biologic free sustained remission at week 24. | week 14 and 24
  Remission achieved and maintained without additional therapy
Need for additional treatment to achieve remission by week 14 | Week 14
  Remission achieved without additional therapy
Mucosal healing as assessed by MRE in dietary responsive disease at week 52 | Week 52
  Mucosal healing

CONTACTS AND LOCATIONS:
Overall Officials: Rotem Sigall Boneh, RD, Principal Investigator — Pediatric Gastroenterology and Nutrition unit; The E. Wolfson.Medical Center; Michal Yaakov, Study Director — Pediatric Gastroenterology and Nutrition unit; The E. Wolfson.Medical Center
Locations (7):
- Canada (3):
  - Dr. Eytan Wine,, Edmonton
  - Johan Van Limbergen, Halifax
  - Dr Sally Lawrence, Vancouver
- Dr. Séamus Hussey, Dublin, Ireland
- The E. Wolfson.Medical Center, Holon, Israel
- Spain (2):
  - Dr. Francisco Javier Martin Carpi, Barcelona
  - Dr. Víctor Manuel Navas López, Málaga

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sigall-Boneh R, Pfeffer-Gik T, Segal I, Zangen T, Boaz M, Levine A. Partial enteral nutrition with a Crohn's disease exclusion diet is effective for induction of remission in children and young adults with Crohn's disease. Inflamm Bowel Dis. 2014 Aug;20(8):1353-60. doi: 10.1097/MIB.0000000000000110. PMID 24983973
- [Background] Levine A, Wine E, Assa A, Sigall Boneh R, Shaoul R, Kori M, Cohen S, Peleg S, Shamaly H, On A, Millman P, Abramas L, Ziv-Baran T, Grant S, Abitbol G, Dunn KA, Bielawski JP, Van Limbergen J. Crohn's Disease Exclusion Diet Plus Partial Enteral Nutrition Induces Sustained Remission in a Randomized Controlled Trial. Gastroenterology. 2019 Aug;157(2):440-450.e8. doi: 10.1053/j.gastro.2019.04.021. Epub 2019 Jun 4. PMID 31170412
- [Background] Sigall Boneh R, Sarbagili Shabat C, Yanai H, Chermesh I, Ben Avraham S, Boaz M, Levine A. Dietary Therapy With the Crohn's Disease Exclusion Diet is a Successful Strategy for Induction of Remission in Children and Adults Failing Biological Therapy. J Crohns Colitis. 2017 Oct 1;11(10):1205-1212. doi: 10.1093/ecco-jcc/jjx071. PMID 28525622
- [Derived] Sigall Boneh R, Navas-Lopez VM, Hussey S, Pujol-Muncunill G, Lawrence S, Rolandsdotter H, Otley A, Martin-de-Carpi J, Abramas L, Herrador-Lopez M, Egea Castillo N, Chen M, Hurley M, Wingate K, Olen O, Eurenius Raaf T, Yaakov M, Wierdsma N, Van Limbergen J, Wine E. Modified Crohn's Disease Exclusion Diet Maintains Remission in Pediatric Crohn's Disease: Randomized Controlled Trial. Clin Gastroenterol Hepatol. 2025 Oct;23(11):2001-2011. doi: 10.1016/j.cgh.2024.12.006. Epub 2024 Dec 26. PMID 39732356